CLINICAL TRIAL: NCT04713527
Title: Polymerase Chain Reaction and Cultivation of the Peritoneal Fluid at Operation for Appendicitis and Postoperative Enteral Antibiotic Treatment. A Feasibility and Non-inferiority Study
Brief Title: Polymerase Chain Reaction (PCR) and Cultivation of the Peritoneal Fluid at Operation for Appendicitis and Postoperative Enteral Antibiotic Treatment
Acronym: PACPAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 115-2019-NQ
Record Dates: First submitted 2020-11-02; First posted 2021-01-19 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-01

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peritoneal Fluid.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cultivation and PCR within 24 hours — During operation for appendicitis peritoneal fluid will be extracted. This is sent to cultivation and PCR analysis to determine if there is bacteria within the peritoneal cavity.
Drug: Enteral antibiotics — Patients with complicated appendicitis will receive enteral antibiotics instead of intravenous

SUMMARY:
Patients diagnosed with acute appendicitis receives antibiotics during the operation, and only patients where the surgeon suspects a complicated appendicitis with spread inflammation to the abdominal cavity receive antibiotics for 3 days postoperative.

In a previous study at the surgical department, the investigators were able to show that the surgeon's assessment during the surgery of whether the appendicitis are complicated or not is very uncertain. This means that some patients receive antibiotics after surgery for no reason, and others might have benefited from antibiotics. The aim of this study is to solve this problem.

By extracting some of the peritoneal fluid, it is possible to investigate whether there are bacteria or not in the abdominal cavity. Today when the fluid is cultivated, the answer will appear after 3-4 days. Therefore a new method is needed which confirms the presence of bacteria in the abdominal cavity within 24 hours.

In this study growth of bacteria in cultivation is examined and determined within 24 hours. The study also want to use PCR analysis. It is a special technique, which examines the fluid from the abdominal cavity for bacteria and provide answer within a few hours. It is investigated whether it is possible to perform this method in the daily routine of the department.

New research also shows that if patients needs antibiotics after surgery they can be treated with tablets instead of injection into the blood vessel. Antibiotic treatment with tablets will mean that the patient can be discharged earlier.

The primary purpose of this study is to investigate whether it is possible with the PCR technique or cultivation to determine whether there are bacteria in the abdominal cavity of patients undergoing surgery for acute appendicitis or not, so that any continued antibiotic treatment after surgery can be targeted to the individual patient. The secondary purpose is to investigate whether antibiotic treatment with tablets are as effective as getting antibiotics into the blood vessel.

The patients participating in the project will undergo the usual routine treatment and surgery. The only exception is retrieval of the naturally occurring fluid from the abdominal cavity. This will be done during the operation by special suction equipment that can be fitted to the usual operating equipment. It will not cause any discomfort or inconvenience to the patient. The technique of extracting fluid from the abdominal cavity has been used in previous studies of patients operated on for acute appendicitis.

The benefit for the patient will be a more targeted antibiotic treatment so that both unnecessary treatment is avoided, and patients who previously would not have received treatment can benefit from this. For society a more targeted antibiotic treatment will mean less risk of developing resistance and less hospitalization.

DETAILED DESCRIPTION:
Aim The primary aim is to investigate whether it is possible to determine if there are bacteria in the patient's peritoneal fluid either from PCR (polymerase chain reaction) or cultivation within 24 hours in patients undergoing surgery for acute appendicitis.

The secondary purpose is to investigate whether oral administered postoperative antibiotic treatment is non-inferior to prior standard intravenous administration therapy focusing on wound infection and intra-abdominal abscess.

The clinical issues

Previous studies from our department have shown that both over- and under treatment with antibiotics in patients operated for acute appendicitis is reality. It has not previously been possible to control the treatment based on the result of peritoneal fluid culture, because the final response to conventional cultivation is first available after a 3-4 days. The PCR (polymerase chain reaction) technique allows diagnostics within hours.

The second problem is that conventional postoperative antibiotic treatment is most often the only reason for the patient to remain hospitalized for at least 3 days. With oral antibiotic treatment the patient can be treated at home.

Hypotheses

* In case of acute appendicitis surgery, it is possible to determine the presence of bacteria in the peritoneal fluid by PCR or culture within 24 hours, and that the final response to D + R after a further 3 days of culture is consistent with this.
* Oral postoperative antibiotic therapy is non-inferior to traditional intravenous administration in complicated appendicitis.

Background Acute appendicitis surgery is one of the most frequent operations with a lifetime risk of approximately 9%.

Appendicitis can be classified as uncomplicated (phlegmonous) or complicated (gangrenous, perforated or peri appendicular abscess) based on perioperative findings. Perioperative antibiotics prophylaxis is administered to all patients, who are operated for acute appendicitis, whether there is complicated or uncomplicated appendicitis due to prevent complications. The complications are primarily wound infection or intra-abdominal abscess. In complicated appendicitis treatment continues for three days after surgery. The antibiotic treatment targets both aerobic and anaerobic intestinal bacteria. Several antibiotic regimens have been found to be equivalent. In our department, cefuroxime and metronidazole as intravenous administration are used as standard.

It is the surgeon who alone determine whether an appendicitis is complicated by the findings under the surgery. A previous study conducted in the ward showed that in 42% of the cases where the surgeon assessed that the appendix was perforated, no bacterial growth could be detected by growing on perioperatively retrieved peritoneal fluid, while in 18% of cases where the histology showed simply phlegmonous appendicitis, there was a positive culture result. Therefore, there is a risk of both under- and over treatment, which is inappropriate for many reasons, including increased resistance development. Therefore, a more evidence-based approach to postoperative antibiotic treatment after surgery for acute appendicitis is needed.

A prerequisite to organize a more appropriate antibiotic treatment will be the ability to obtain a reliable culture result from peritoneal fluid within 24 hours. Conventional cultivation can be problematic because not all bacteria will show growth within this time. PCR could be a better method and an alternative to ordinary culture.

If it is found that it is possible within 24 hours after the operation to determine whether there is growth of bacteria in the peritoneal fluid, it will be possible to let this determine if continued postoperative treatment are needed regardless of the operative findings, thus reducing the risk of under- or overtreatment.

Another important clinical question is whether antibiotics should be given intravenous or oral. Oral treatment will be convenient for both the patient and the health care system, as the patient will then be able to be treated at home. A previous retrospective Danish study has shown that oral antibiotic treatment is equivalent to intravenous treatment and that the hospitalization time can be reduced by an average of 61 hours. Oral treatment has been introduced in some Danish hospitals.

Method The study design is a prospective cohort/feasibility and non-inferior study, which includes a total of 100 patients older than 18 who undergo an appendectomy due to acute appendicitis.

When diagnostic laparoscopy is performed and appendicitis is recognized, 10 ml of peritoneal fluid is extracted for examination by special equipment approved for this purpose. In the absence of peritoneal fluid, the surgeon will rinse with 20 ml of sterile saline corresponding to the peri appendicular area. The peritoneal fluid is then sent for PCR, culture and resistance determination.

When these procedures are performed usual antibiotic treatment in the form of 3 g of cefuroxime and 1.5 g of metronidazole are administered intravenously and the operation is performed according to usual guidelines.

If there is a complicated appendicitis (assessed preoperatively), oral antibiotic treatment in the form of 875 mg amoxicillin / 125mg clavulanic acid + 500mg metronidazole x 3 daily for 3 days are prescribed. The treatment will be independent to the result of PCR determination and the culture on the peritoneal fluid.

The sample containing the peritoneal fluid is sent to the microbiological department, where they make the cultivation and resistance determination as well as the PCR. Growth is observed on the cultures at 12, 24 and 36 hours and the final result with resistance determination after 3 days. The type of bacteria in the samples are recorded. Follow-up is done 30 days postoperative, where the patient is contacted by telephone for postoperative complications. Complications for appendicitis are typically intraabdominal abscess and wound infection, and therefore special attention will be given to these. Wound infections are defined by the Centers for Disease Control and Prevention (CDC) surgical site infections (SSI). These and any other complications are also recorded according to the Clavien Dindo classification (CD).

The part of the study that deals with the PCR and culture on the peritoneal fluid is a descriptive study to investigate whether the PCR technique can be introduced into the daily clinic. The technique has not previously been tested anywhere and therefore it is not possible to make any strength calculation on the sensitivity and specificity of the PCR method relative to the result of the final culture. From our previous studies it is known that at least one third of the patients will be classified as having a complicated appendicitis. The inclusion of 100 patients will in our opinion be enough to be able to calculate sensitivity and specificity with acceptable safety limits, which can be indicative of further studies.

The other part of the study concerns the change of antibiotic treatment from intravenous to oral treatment. The basis for assessing this will be the frequency of any infectious complications compared to the frequencies present in the literature. Wound infections by the laparoscopic technique is about 3% and intra-abdominal abscess is about 7.5%. The investigators will continuously record the frequency of these complications, and if deviations from the above occur a detailed review of each case will be made and a decision on whether this part of the project can continue or not. The results will also be indicative of whether a randomized trial will be necessary.

Project feasibility All methods are tested. The method of taken samples from the peritoneal fluid is tested in another study at the department. The study itself is a feasibility study to see if it is safe and possible to use these methods in the clinic. For these reasons, a pilot study is not necessary.

Limitation The exclusion criteria are a limitation. Especially the age limit of 18 years courses that the generalizability to patients under 18 is not possible. It is a problem because there is a lot of patients with appendicitis under the age of 18.

It is also a limitation that the study only includes 100 patients. The reason for this is that the study is a feasibility study and therefore believed 100 patients is enough to conclude if further studies are needed.

Expected clinical impact The results could be of great importance for future treatment. If it is possible to get an answer of the presence of bacteria in the peritoneal fluid within 24 hours, it is possible to target the antibiotic treatment to the right patients. This is important for the single patient but also important for the society because the use of antibiotic leads to development of antibiotic resistant bacteria and therefore it is important to avoid unnecessary use of antibiotic. Since appendicitis is a very frequent disease, research in this area is of great importance as it involves a high number of patients and thus a large amount of antibiotics. Especially because it is shown that the surgeons overestimate the number of patients with complicated appendicitis.

In addition to this the oral treatment has the impact that most patients can be treated with antibiotics at home. This will have a positive impact for both patient and society.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing diagnostic laparoscopy with suspected acute appendicitis
* Admitted by the Emergency Department (FAM), at Odense University Hospital (OUH) or Svendborg
* Gets a laparoscopic appendectomy.
* Speaks and understands Danish

Exclusion Criteria:

* Age under 18
* Pregnant or breastfeeding
* Language difficulties
* Sepsis preoperatively assessed via the SIRS criteria leading to preoperatively administered antibiotics.
* Patients with known gastrointestinal disorders as chronic inflammatory bowel disease or previous cancer disease.
* Open appendectomy
* Other illness than acute appendicitis

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Admitted by the Emergency Department (FAM), at OUH or Svendborg
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-05-29 (Estimated); Study Completion 2021-06-28 (Estimated)

PRIMARY OUTCOMES:
Cultivation answer within 24 hours | 24 hours after surgery
  A sample of peritoneal fluid is observed for growth of bacteria in Department of Clinical Microbiology within 24 hours after surgery. The answer is either positive (growth of bacteria) or negative (no growth of bacteria).
PCR answer within 24 hours | 24 hours after surgery
  A sample of peritoneal fluid is analysed with the PCR-method. The outcome is either positive (detection of bacterial DNA) or negative (no detection of bacterial DNA)
Complications | 30 days follow up
  Wound infection, intraabdominal abscess and other

SECONDARY OUTCOMES:
Descriptive data - sex | 1 day
  Female or male is registred. Data is collected from the patients personal journal.
Descriptive data - height | 1 day
  The patients height in centimeters is registred. Data is collected from the patients personal journal.
Descrriptive data - weight | 1 day
  The patients weight in kilograms are registred. Data is collected from the patients personal journal.
Descriptive data - American Society of Anesthesiologists (ASA) score | 1 day
  ASA I: A normal healthy patient ASA II: A patient with mild systemic disease ASA III: A patient with severe systemic disease ASA IV: A patient with severe systemic disease that is a constant threat to life ASA V: Moribund patinet who is not expected to survive without the operation Data is collected from the patients personal journal.
Descriptive data - smoking status | 1 day
  It is registred if the patient is a smoker, former smoker or non-smoker. Also packages years are calculated. Data is collected from the patients personal journal.
Descrptive data - alcohol status | 1 day
  It is registred if the patients drinks more alcohol items a week than 7 items for women and 14 items for men. Data is collected from the patients personal journal.
Descriptive data - Systemic Inflammatoric Response Syndrome (SIRS) criteria | 1 day
  SIRS is defined as fulfilling at least two of the following four criteria: fever >38.0°C or hypothermia <36.0°C, tachycardia >90 beats/minute, tachypnea >20 breaths/minute, leucocytosis >12*109/l or leucopoenia <4*109/l. Data is collected from the patients personal journal.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, OUH, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhangu A, Soreide K, Di Saverio S, Assarsson JH, Drake FT. Acute appendicitis: modern understanding of pathogenesis, diagnosis, and management. Lancet. 2015 Sep 26;386(10000):1278-1287. doi: 10.1016/S0140-6736(15)00275-5. PMID 26460662
- [Background] Daskalakis K, Juhlin C, Pahlman L. The use of pre- or postoperative antibiotics in surgery for appendicitis: a systematic review. Scand J Surg. 2014 Mar;103(1):14-20. doi: 10.1177/1457496913497433. Epub 2013 Sep 20. PMID 24056131
- [Background] van Rossem CC, Schreinemacher MH, Treskes K, van Hogezand RM, van Geloven AA. Duration of antibiotic treatment after appendicectomy for acute complicated appendicitis. Br J Surg. 2014 May;101(6):715-9. doi: 10.1002/bjs.9481. Epub 2014 Mar 26. PMID 24668341
- [Background] Tind S, Qvist N. Acute Appendicitis: A Weak Concordance Between Perioperative Diagnosis, Pathology and Peritoneal Fluid Cultivation. World J Surg. 2017 Jan;41(1):70-74. doi: 10.1007/s00268-016-3686-8. PMID 27541029
- [Background] Kleif J, Rasmussen L, Fonnes S, Tibaek P, Daoud A, Lund H, Gogenur I. Enteral Antibiotics are Non-inferior to Intravenous Antibiotics After Complicated Appendicitis in Adults: A Retrospective Multicentre Non-inferiority Study. World J Surg. 2017 Nov;41(11):2706-2714. doi: 10.1007/s00268-017-4076-6. PMID 28600695
- [Background] National Collaborating Centre for Women's and Children's Health (UK). Surgical Site Infection: Prevention and Treatment of Surgical Site Infection. London: RCOG Press; 2008 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK53731/ PMID 21698848
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542